CLINICAL TRIAL: NCT04810897
Title: Effects of Home-based Exercise Programme in Individuals With Parkinson's Disease
Brief Title: Effects of Home-based Exercise in Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-CIRB 2020/048.1902
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: Exercise; Gait characteristics
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease: The neurologists will inform the individuals with PD that we are doing this research and we will attach the research advertisement at Movement Disorder Clinic, Division of Neurology, Faculty of Medicine Siriraj Hospital, Mahidol University, Thailand. Only individuals with PD who meet the inclusion and exclusion criteria will be invited to participate in the study. The researcher will inform participants about the purpose, procedure, and advantage of the study prior to participation in the study. Individuals with PD will be asked to sign an informed consent if they agree to participate in the study.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise programme is reported in the clinical trial registration number is NCT03473834.

SUMMARY:
Home-based exercise program focusing on axial rigidity could be used as an adjunct rehabilitation program to improve rotational movement, gait and functional movement associated with axial rigidity in individuals with PD.

DETAILED DESCRIPTION:
Typically, individuals with PD revert to more primitive movement patterns, which lack many of the automatic postural adjustments and axial movements that accompany simple activities, such as supine to standing, getting up from sitting or turning over in bed. The present study is designed to allow patients and their relatives to perform exercises by themselves conveniently at home. The results were considered a vital component of a complex intervention and were played an integral part in the implementation process of exercises in functional performance. Furthermore, this study will prove sufficient high-quality evidence to investigate whether improvements in function due to exercise-based rehabilitation are associated with reducing axial rigidity in individuals with PD.

Currently, there is a lack of evidence for the effectiveness of home-based exercise programs in PD patients in Thailand. For the present study, we devised a home-based 10-week exercise program focusing on segmental rotation and task-specific movements for turning practice to determine effects on axial mobility and turning. The aimed of this study to examine the effects of a 10-week task specific home-based exercise program on turning kinematics, gait and stepping characteristics, the Functional Reach test (FRT), the Unified Parkinson's Disease Rating Scale (UPDRS), the Freezing of Gait questionnaire (FOG) and the Fall Efficacy Scale International (FES-I) in individuals with PD.

ELIGIBILITY:
1. Inclusion Criteria;

   * Clinically diagnosed with PD stages 1.5 to 3 as assessed by the modified Hoehn and Yahr scale
   * The age groups between 50 and 75 years
   * Taking PD medication regularly for at least a month
   * No signs of wearing-off phenomenon
   * Able to walk independently without any assistive device and 6) able to follow commands and instructions
2. Exclusion Criteria;

   * Clinically diagnosed with dementia or other neurological or cardiopulmonary diseases
   * Musculoskeletal problems that could influence the test performance such as arthritis or severe leg pain
   * High blood pressure (more than 140/90 mmHg)
   * Haemodialysis
   * Visual problems that could not be adjusted with lenses or glasses
   * Taking medicine which affected to functional movement.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with Parkinson's disease (PD) who refers from a public hospital and recruits from community.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
The Unified Parkinson's Disease Rating Scale (UPDRS), | 3 months
  The UPDRS consists of four major parts: 1) mental, behavior and mood, 2) activities of daily living, 3) motor examination and 4) complications of therapy, in totally 42 items. Each item has multiple points that include zero for normal or no problems, 1 for minimal problems, 2 for mild problems, 3 for moderate problems and 4 for severe problems. The higher score would indicate the more severe problems in individuals with PD.
Functional axial rotation - physical (FAR) | 3 months
  A clinical measurement for axial mobility, which is usually used to measure spinal flexibility. If the FAR yields a high score, it implies better flexibility, axial movement and postural control and balance.
Gait and turning characteristics | 3 months
  Gait will be measure by the participants will stand at the edge of the platform (The Zebris FDM-System-Gait Analysis; Zebris Medical GmbH, Isny, Germany) and will be asked to walk barefoot at a comfortable speed to the other end of the platform, this will be repeated for a total of 3 trials. The averaged data including foot rotation (deg), step width (cm), step length (cm), step time (sec), cadence (steps/min) and gait velocity (km/s) were analysed and used in the comparisons. Turning kinematics (the onset latencies of body segments reorientation and stepping characteristics) will be recorded during participants performed a turning on level ground at 180° in standing position by using the Inertial Measurement Unit (xIMU) (x-IMU, x-io Technologies Ltd., UK).

SECONDARY OUTCOMES:
Time Up and Go | 3 months
  The average of 3 attempts of the time required to rise from a chair, walk 3 m, return to the chair, and sit down again will be collected. The faster times indicate better balance and mobility.
10 Meter walk test | 3 months
  Participants will be instructed to walk at a comfortable pace following a 10-meter distance marked on the floor. The time of 10 Meter walk test will be calculated
Global rating scale (GROC) | 3 months
  A GROC score of zero will be considered as unchanged, and GROC scores of +1, +2, +3, +4 and +5 represent an increase in perceived improvement. In contrast, GROC scores of -1, -2, -3, -4, and -5 indicate the degree of perceived deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Fuengfa Khobkhun, Principal Investigator — Physical Therapy
Locations (1):
- Fuengfa Khobkhun, Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No
Data from the patients so, it could be privacy to ask for IPD data.